CLINICAL TRIAL: NCT03298503
Title: Effects of Task Prioritization on Postural-suprapostural Task and Brain Activity in Parkinson's Disease With Different Balance Ability: During Standing and Walking
Brief Title: Task-priority Effects on Postural-suprapostural Task in Patients With Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 201701080RINB
Record Dates: First submitted 2017-05-04; First posted 2017-10-02 (Actual); Last update posted 2018-01-02 (Actual); Status verified 2017-05

CONDITIONS: Parkinson Disease
Keywords: Parkinson's disease; posture balance; attention
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- early stage or non-freezers PD (Active Comparator): early stage defined as modified Hoehn and Yahr scale 1, 1.5 and 2, means that symptoms involved unilateral or bilateral without impairment of balance.
  non-freezers defined as without freezing of gait, means that patients without transient inability to generate effective stepping.
  Interventions: Other: task-priority strategies
- moderate stage or freezers PD (Experimental): moderate stage defined as modified Hoehn and Yahr scale 2.5 and 3, means that symptoms involved unilateral or bilateral without impairment of balance.
  freezers defined as with freezing of gait, means that patients have transient inability to generate effective stepping.
  Interventions: Other: task-priority strategies

INTERVENTIONS:
Other: task-priority strategies — posture-focus strategy: when performing postural-suprapostural task (dual-task), the patient mainly focus on postural task (standing/walking).
  supraposture-focus strategy: when performing postural-suprapostural task (dual-task), the patient mainly focus on suprapostural task (stabilize the tray).

SUMMARY:
Postural-suprapostural task is defined as postural control takes place while at least one other concurrent task is being performed. In a postural-suprapostural task, appropriate prioritization of is necessary to achieve task goals and maintain postural stability. Therefore, regarding to impose task prioritization in a postural-suprapostural task, the optimal task-priority strategy for PD patients is still an issue of debate. With the uses of EEG, EMG and behavioral measures, the purpose of this project is to investigate the differences in performance quality and intrinsic neural mechanisms of a postural-suprapostural task for PD patients, by adopting posture-focus and suprapostural-focus strategies during standing and walking. The present project is expected to have significant contributions not only to gain a better insight to neural correlates of concurrent postural and suprapostural tasks with different task prioritization under standing and walking, but to optimize treatment strategy for PD patients with balance or dual-tasking disturbances.

DETAILED DESCRIPTION:
Postural-suprapostural task is defined as postural control takes place while at least one other concurrent task is being performed. In a postural-suprapostural task, appropriate prioritization of is necessary to achieve task goals and maintain postural stability. Some studies support that a "posture-first" strategy is favored by patients with Parkinson disease (PD) in order to secure stance stability, but this comes at the cost of reduced suprapostural performance. In addition, overemphasizing on postural task might deteriorate automatic control of posture resulting in increased postural instability, and the best task-priority strategy might vary with balance ability of PD patients. Therefore, regarding to impose task prioritization in a postural-suprapostural task, the optimal task-priority strategy for PD patients is still an issue of debate. With the uses of EEG, EMG and behavioral measures, the purpose of this 2-year research project is to investigate the differences in performance quality and intrinsic neural mechanisms of a postural-suprapostural task for PD patients, by adopting posture-focus and suprapostural-focus strategies during standing and walking. In the first year, we will characterize task prioritization effect on reciprocity of a postural-suprapostural task, with a special focus on modulation of brain and muscle activity patterns in standing posture for early stage (modified H & Y: 1, 1.5 and 2) and moderate stage (modified H & Y: 2.5 and 3) PD patients. In the second year, the appropriate task prioritization, walking automaticity and power/connectivity of brain areas will be investigated in walking for PD patients with/without freezing of gait. The present project is expected to have significant contributions not only to gain a better insight to neural correlates of concurrent postural and suprapostural tasks with different task prioritization under standing and walking, but to optimize treatment strategy for PD patients with balance or dual-tasking disturbances.

ELIGIBILITY:
inclusion criteria:

1. patients with Parkinson's Disease in H&Y stage from stage 1 to stage 3
2. without other neurological disease with balance impairment
3. can stand and walk without aids for at least 30 seconds

exclusion criteria:

1. Mini-Mental State Examination > 27
2. Questionnaire for Impulsive-Compulsive Disorders in Parkinson's Disease-Rating Scale (QUIP-RS) < 10
3. Hamilton Depression Rating Scale (HAM-D) < 17
4. pregnancy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-12-05 (Actual); Primary Completion 2017-12-05 (Actual); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Electroencephalography (EEG) | about 30 seconds for each trial, total about 30 minutes
  to collect the brain activity (unit: uV)
Electromyography (EMG) | about 30 seconds for each trial, total about 30 minutes
  to collect the muscle activity (unit: mV)

SECONDARY OUTCOMES:
Gait parameters (GAITRite) | about 30 seconds for each trial, total about 30 minutes
  to know how the subjects walk during the trial
Center of pressure (COP) | about 30 seconds for each trial, total about 30 minutes
  to know how the subjects stand during the trial
Tilting angle of inclinometer | about 30 seconds for each trial, total about 30 minutes
  to know how the subjects perform the suprapostural task during the trial

CONTACTS AND LOCATIONS:
Overall Officials: Cheng-Ya Huang, Ph.D., Principal Investigator — School & Graduate Institute of Physical Therapy, College of Medicine, National Taiwan University
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Peterson DS, Fling BW, Mancini M, Cohen RG, Nutt JG, Horak FB. Dual-task interference and brain structural connectivity in people with Parkinson's disease who freeze. J Neurol Neurosurg Psychiatry. 2015 Jul;86(7):786-92. doi: 10.1136/jnnp-2014-308840. Epub 2014 Sep 15. PMID 25224677
- [Background] Kelly VE, Eusterbrock AJ, Shumway-Cook A. A review of dual-task walking deficits in people with Parkinson's disease: motor and cognitive contributions, mechanisms, and clinical implications. Parkinsons Dis. 2012;2012:918719. doi: 10.1155/2012/918719. Epub 2011 Oct 27. PMID 22135764
- [Background] Shumway-Cook A, Woollacott M, Kerns KA, Baldwin M. The effects of two types of cognitive tasks on postural stability in older adults with and without a history of falls. J Gerontol A Biol Sci Med Sci. 1997 Jul;52(4):M232-40. doi: 10.1093/gerona/52a.4.m232. PMID 9224435
- [Background] Beck EN, Ehgoetz Martens KA, Almeida QJ. Freezing of Gait in Parkinson's Disease: An Overload Problem? PLoS One. 2015 Dec 17;10(12):e0144986. doi: 10.1371/journal.pone.0144986. eCollection 2015. PMID 26678262
- [Background] Mitra S, Fraizer EV. Effects of explicit sway-minimization on postural--suprapostural dual-task performance. Hum Mov Sci. 2004 Jun;23(1):1-20. doi: 10.1016/j.humov.2004.03.003. PMID 15201038
- [Background] Vervoort G, Heremans E, Bengevoord A, Strouwen C, Nackaerts E, Vandenberghe W, Nieuwboer A. Dual-task-related neural connectivity changes in patients with Parkinson' disease. Neuroscience. 2016 Mar 11;317:36-46. doi: 10.1016/j.neuroscience.2015.12.056. Epub 2016 Jan 5. PMID 26762801
- [Background] Knaepen K, Mierau A, Tellez HF, Lefeber D, Meeusen R. Temporal and spatial organization of gait-related electrocortical potentials. Neurosci Lett. 2015 Jul 10;599:75-80. doi: 10.1016/j.neulet.2015.05.036. Epub 2015 May 21. PMID 26003448
- [Derived] Huang CY, Chen YA, Wu RM, Hwang IS. Neural Oscillations and Functional Significances for Prioritizing Dual-Task Walking in Parkinson's Disease. J Parkinsons Dis. 2024;14(2):283-296. doi: 10.3233/JPD-230245. PMID 38457151
- [Derived] Hung YT, Chen LC, Wu RM, Huang CY. The Effects of Task Prioritization on Dual-Tasking Postural Control in Patients With Parkinson Disease Who Have Different Postural Impairments. Arch Phys Med Rehabil. 2020 Jul;101(7):1212-1219. doi: 10.1016/j.apmr.2020.02.014. Epub 2020 Mar 28. PMID 32234414